CLINICAL TRIAL: NCT01280292
Title: Central Hypothyroidism,a New Laboratory Approach for Hormone Measurement
Brief Title: Central Hypothyroidism, a Novel Laboratory Measurement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Ruth Percik M.D., Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SHEBA-10-8213-RP-CTIL
Record Dates: First submitted 2011-01-19; First posted 2011-01-20 (Estimated); Last update posted 2011-02-03 (Estimated); Status verified 2011-02

CONDITIONS: Central Hypothyroidism
Keywords: central hypothyroidism, hypopituitarism, eltroxin
MeSH Terms: conditions — Hypothyroidism; Hypopituitarism | interventions — Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Eltroxin — Eltroxin dosage titration according to free T4 measurement every 3 months

SUMMARY:
Medical management of central hypothyroidism is controversial due to lack of reference for evaluation of pituitary negative feedback. Therefore, titration of medical treatment is based on T4 levels, measured with variable laboratory methods. Patients who have central hypothyroidism usually have concomitant deficiencies in other pituitary hormones for which they need replacement therapy such as steroids, testosterone and growth hormone. This combined hormone deficiency makes clinical and laboratory evaluation challenging among these patients. Symptomatically, central hypothyroidism is relatively mild and lack non-specific and it might be overlooked due to other hormonal deficiencies. Replacement therapy for central hypothyroidism is titrated by arbitrary target free T4 levels of above 50th percentile of normal. The goal of our study is to compare the standard results from well known measure methods to a new method for measuring Ft4 using Liquid chromatography - tandem mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* Clinical evidence of central hypothyroidism: status post pituitary surgery and/or radiotherapy plus laboratory documentation of central hypothyroidism, with or without concurrent hormonal deficiencies in other axes, such as ACTH, LH, FSH

Exclusion Criteria:

* Primary hypothyroidism

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-02 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
free T4 levels | a year

SECONDARY OUTCOMES:
Symptoms of hypothyroidism | a year

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Percik, M.D., Principal Investigator — Sheba Medical Center